CLINICAL TRIAL: NCT04692272
Title: Effects of Xbox Kinect Exercise Training on the Sleep Quality, Anxiety and Functional Capacity in Older Adults
Brief Title: Xbox Kinect, Sleep Quality, Anxiety and Functional Capacity in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giselle Soares Passos, Associate Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.040.278
Record Dates: First submitted 2020-12-24; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Sleep; Anxiety; Aging; Exercise
MeSH Terms: conditions — Anxiety Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL group (No Intervention): The CONTROL group did not exercise.
- XBOX group (Experimental): The XBOX group performed exercise for 60 min, three times/week, for 6 weeks, using the Xbox Kinect game "Your Shape Fitness evolved". This game was chosen because it simulates an environment with a variety of physical activities, in which the majority can be practiced by older adults. The activities were carried out individually. The game activities selected for the physical activity sessions were: 1) Zen-Develop it (stretching, balance and flexibility activities, similar to Yoga); 2) Pump it (to fill balls until they burst); 3) Wall Breaker (to break blocks, similar to boxing); 4) Kick it (soccer activity); 5) Hurricane (to lift the balls off the floor and not let them fall); 6) Stack in Up (balance activity).
  Interventions: Behavioral: Exercise in the XBOX kinect

INTERVENTIONS:
Behavioral: Exercise in the XBOX kinect — The XBOX group performed exercise for 60 min, three times/week, for 6 weeks, using the Xbox Kinect game "Your Shape Fitness evolved". This game was chosen because it simulates an environment with a variety of physical activities, in which the majority can be practiced by older adults. The activities were carried out individually. The game activities selected for the physical activity sessions were: 1) Zen-Develop it (stretching, balance and flexibility activities, similar to Yoga); 2) Pump it (to fill balls until they burst); 3) Wall Breaker (to break blocks, similar to boxing); 4) Kick it (soccer activity); 5) Hurricane (to lift the balls off the floor and not let them fall); 6) Stack in Up (balance activity).
  Arms: XBOX group

SUMMARY:
The present study aims to examine the effects of Xbox Kinect exercise training program on the sleep quality, anxiety and functional capacity in older adults. Older adults were randomized into two groups. The XBOX group performed exercise with Xbox Kinect during 60 min, three times/week for 6 weeks. The CONTROL group did not exercise. Pittsburgh Sleep Quality Index was used to evaluate sleep quality, anxiety symptoms by the State-Trait Anxiety Inventory, and the functional capacity was analyzed using following tests: Chair Stand Test, 8-Foot Up and Go Test, and 6-min Walk Test.

ELIGIBILITY:
Inclusion Criteria:

1. ability to perform exercises with Xbox Kinect and/or physical/functional tests and to answer the questionnaires;
2. score ≥ 24 on the Mini-Mental State Examination

Exclusion Criteria:

(a) using psychiatric drugs or beta-blockers;

1. functional limitations
2. exercise regularly

(e) smoking (b) previous experience with Xbox Kinect games.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2015-02-15 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Sleep Quality at 6 weeks | up to 24 weeks
  Sleep Quality: Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month time interval and provides quantitative and qualitative information on sleep. The questionnaire consists of 19 self-report items and other questions. The score ranges from 0 to 21 and scores > 5 indicates the patient is a poor sleeper

SECONDARY OUTCOMES:
Change from Baseline Anxiety at 6 weeks | up to 24 weeks
  Anxiety Symptoms: State-Trait Anxiety Inventory (STAI) assesses anxiety level using two scales (State and Trait) with 20 items. Range of scores is 20-80, and the scores indicate low (0-30), medium (31-49), or high (50 or more) anxiety levels
Change from Baseline strength at 6 weeks | up to 24 weeks
  Chair Stand Test is used to assess lower body strength. After a signal participants completed as many "stand-ups" as possible with 30s. Total repetitions completed within 30s are used to score the participants' performance.
Change from Baseline agility/dynamic balance at 6 weeks | up to 24 weeks
  The 8-ft Timed Up & Go Test is used to assess agility and dynamic balance. Participants are asked to sit on a chair. On cue, they stood up, walked as quickly as possible around a cone set 8ft from the chair, and sat back down on the chair. Total time to complete the test in seconds was measured to assess performance.
Change from Baseline aerobic endurance at 6 weeks | up to 24 weeks
  The 6-MWT is performed in a 20-m-long indoor hallway free of obstacles. Participants are instructed to walk at a self-selected regular pace to cover as much distance as they could during the allotted time. The score is the total number of meters walked in 6 min

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evangelista de Lima B, Passos GS, Youngstedt SD, Bandeira Santos Junior LC, Goncalves Santana M. Effects of Xbox Kinect exercise training on sleep quality, anxiety and functional capacity in older adults. J Bodyw Mov Ther. 2021 Oct;28:271-275. doi: 10.1016/j.jbmt.2021.07.029. Epub 2021 Aug 6. PMID 34776152